CLINICAL TRIAL: NCT00132561
Title: A Double-blind, Randomised, Placebo-controlled Trial to Measure the Potential of Intermittent Treatment With Artesunate Plus Sulphadoxine/Pyrimethamine (SP) to Reduce the Malaria Burden in Sub-Saharan Africa
Brief Title: A Trial of Intermittent Treatment in the Prevention of Malaria in Senegalese Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Institut de Recherche pour le Developpement, Senegal (Other); Institut de Recherche pour le Developpement (Other Government); Cheikh Anta Diop University, Senegal (Other); Ministry of Health, Senegal (Other Government)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: ITCR 5094
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — sulfadoxine-pyrimethamine-artesunate

INTERVENTIONS:
Drug: Sulfadoxine/pyrimethamine and artesunate

SUMMARY:
In countries of the Sahel and sub-Sahel, malaria transmission is highly seasonal with nearly all infections occurring during a few months of the year. However, mortality and morbidity from malaria may be high during this period, especially in young children who are the group most at risk.

Intermittent preventative treatment (IPT) is a new approach to the prevention of malaria in this situation. IPT involves the administration of an anti-malarial to children at risk for malaria at fixed times, even if they are not infected. To investigate how effective this approach might be in Senegal, a trial has been undertaken in which 1136 children aged 6 weeks to 59 months were given a single dose of sulfadoxine pyrimethamine and artesunate on three occasions during a three-month rainy season and the incidence of clinical malaria in these children was compared with that in a group of children who received placebo. Additional observations were made on the incidence of side effects in children in the two groups and on the impact of IPT in children (IPTc) on markers of drug resistance in children whose blood films were positive for Plasmodium falciparum.

DETAILED DESCRIPTION:
Background:

In countries of the Sahel and sub-Sahel, malaria transmission is highly seasonal. Nevertheless, mortality and morbidity from malaria may be very high during the few months of the year when malaria transmission takes place, especially in children. It has been shown previously in The Gambia and elsewhere that in areas of seasonal malaria transmission, mortality and morbidity from malaria in children can be reduced substantially by the regular administration of anti-malarial drugs during the period of risk (chemoprophylaxis). However, chemoprophylaxis is difficult to sustain. Intermittent preventative treatment (IPT) is an adapted form of chemoprophylaxis in which anti-malarial drugs are given at fixed but less frequent intervals than with chemoprophylaxis, allowing blood concentrations of anti-malarial drugs to fall below the inhibitory concentration for periods between drug administrations. This approach to malaria control was used first in pregnant women among whom it is highly effective. However, more recently, it has also been used in infants (IPTi) with anti-malarials being given at the same time as vaccines are administered. This approach is likely to be most effective in areas of high transmission where a high proportion of severe cases of malaria occur in children during the first year of life. IPTi is likely to be less effective in reducing the burden of malaria in areas of seasonal malaria transmission where many cases of severe malaria occur in older children. Intermittent preventative treatment in children (IPTc) is a possible approach to the control of malaria in areas where the main burden of malaria is in older children. Thus, the investigators have undertaken a study to determine how effective this approach would be in preventing malaria in Senegal.

Objectives:

The primary objective of the study was to determine whether the administration of one dose of sulfadoxine-pyrimethamine plus artesunate to Senegalese children aged 6 weeks to 59 months on three occasions during the malaria transmission season would reduce significantly the incidence of clinical attacks of malaria. Secondary objectives were determination of the incidence of side effects in children who received IPTc; the impact of IPTc on the prevalence of molecular markers of resistance to SP in samples positive for Plasmodium falciparum; and the effects of IPTc on the incidence of malaria in the rainy season following the intervention.

Study Area:

The study was conducted in Niakhar, a rural area in the centre of Senegal where malaria transmission is very seasonal, nearly all transmission taking place during a three to four month period. The entomological inoculation rate in the area is about 10 infectious bites per person per year.

Study Population:

All children aged 6 weeks to 59 months residing in the study area were eligible to join the study. There were few exclusion criteria (see below).

Study Procedure:

A series of meetings were held with members of the communities where the trial was undertaken to explain its purpose. The families of potentially eligible children were visited and asked if they wished their child to join the trial. If this was the case, informed consent was obtained. Children were then allocated to one of eight randomisation groups (four active drugs and four placebo).

At the start of the malaria transmission season, all study children were examined and a finger-prick blood sample obtained for determination of packed cell volume and for preparation of a thick blood film for microscopy. A drop of blood was collected onto filter paper and stored for subsequent molecular studies. Children who were anaemic were treated. A similar survey was conducted at the end of the malaria transmission season.

Following initial evaluation children were treated with either a single dose of sulfadoxine-pyrimethamine and artesunate or with matching placebos. Treatment was repeated on two further occasions separated by a period of a month. After each round of drug administration a randomly selected group of children were visited and their parents or guardians asked about any side effects related to the drug administration.

Surveillance for clinical attacks of malaria was undertaken through the detection of study children when they presented to one of the clinics in the study area for treatment of a febrile illness and through weekly home visits.

In the year following the treatment trial, children who had been randomised previously to receive active drug or placebo were followed for another rainy season and the occurrence of clinical attacks malaria detected as described above.

Blood films were stained with Giemsa and examined for malaria parasites by two experienced microscopists. Parasite DNA was extracted from filter paper samples of children who were parasitaemic and examined for mutations in the dhfr and dhps genes associated with resistance to pyrimethamine and to sulphonamides respectively.

Trial End-Points:

The primary trial end-point was the incidence of clinical attacks of malaria in children who received IPTc or placebo. Clinical malaria was defined as an episode of fever (temperature recorded to be 37.5 degrees Celsius or higher or a history of fever within the previous 24 hours) for which no other cause could be found and the presences of P. falciparum parasitaemia at a density of 3,000 parasites per microlitre or greater. This parasite density was chosen as it has been shown previously to be an appropriate fever threshold in the study area. Secondary end-points included the incidence of side effects in children in each group, changes in the prevalences of resistance markers and the incidence of clinical malaria in the year following the main trial.

Sample Size:

It was assumed on the basis of previous information that children in the control group would experience an average of 0.4 clinical attacks of malaria during the malaria transmission season. On the basis of this assumption, a trial with 540 children in each arm would have 80% power at the 5% level of significance to detect a 30% reduction in the incidence of clinical attacks of malaria and a 90% power to detect a 40% reduction including an allowance for a 10% drop-out during the surveillance period.

Monitoring:

The trial was monitored by an independent Data, Safety and Monitoring Board which reviewed the study protocol, the standard operating procedures and the analytical plan.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6 weeks to 59 months
* Residence in the study area
* Informed consent

Exclusion Criteria:

* Known allergy to study drugs
* Serious underlying illness

Ages: 6 Weeks to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200
Dates: Start 2002-06; Study Completion 2003-12

PRIMARY OUTCOMES:
Clinical episodes of malaria

SECONDARY OUTCOMES:
Side effects
Change in the prevalence of drug resistance markers

CONTACTS AND LOCATIONS:
Overall Officials: Badara Cisse, MD, Principal Investigator — Institut de Recherche pour le Developpement, Senegal
Locations (1):
- Institut de recherche pour le developpement, Dakar, Senegal

REFERENCES:
- [Result] Cisse B, Sokhna C, Boulanger D, Milet J, Ba el H, Richardson K, Hallett R, Sutherland C, Simondon K, Simondon F, Alexander N, Gaye O, Targett G, Lines J, Greenwood B, Trape JF. Seasonal intermittent preventive treatment with artesunate and sulfadoxine-pyrimethamine for prevention of malaria in Senegalese children: a randomised, placebo-controlled, double-blind trial. Lancet. 2006 Feb 25;367(9511):659-67. doi: 10.1016/S0140-6736(06)68264-0. PMID 16503464